CLINICAL TRIAL: NCT02393963
Title: Role of Low Dose Intra-articular Tranexamic Acid in the Reduction of Blood Transfusions in Primary Total Hip and Total Knee Arthroplasty: A Randomized Placebo Controlled Study
Brief Title: Intra-articular Tranexamic Acid in the Reduction of Blood Transfusions in Primary Total Hip and Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orthopaedic Innovation Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B2013-089
Record Dates: First submitted 2015-03-03; First posted 2015-03-20 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2016-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (Experimental): Intra-articular administration of low dose Tranexamic acid
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Sodium Chloride
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — 0.5g Tranexamic Acid in 0.9% Sodium Chloride (study group) will be injected into the joint after final closure through a temporary catheter that is brought out through the incision.
  Other Names: DIN#: 02246365, Sandoz Canada Inc.
  Arms: Tranexamic Acid
Other: Placebo — 0.9% Sodium Chloride (placebo group) will be injected into the joint after final closure through a temporary catheter that is brought out through the incision.
  Other Names: Sodium Chloride solution
  Arms: Placebo

SUMMARY:
This is a randomized, double blinded, controlled trial in patients undergoing elective Total Knee Arthroplasty (TKA) and Total Hip Arthroplasty (THA). The study group will receive intra-articular Tranexamic Acid (TXA) while the control group will receive normal saline placebo.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine if intra-articular administration of low dose TXA following THA and TKA results in a clinically relevant reduction in blood loss. The secondary purpose is to determine if there is an increased risk of thromboembolic phenomena with the use of TXA following elective THA and TKA. The primary outcome metric will be - drop in hemoglobin following surgery; secondary metrics include blood loss, transfusion rate, d-dimers, troponin levels, symptomatic deep venous thrombosis (DVT) and pulmonary embolism (PE), vascular events (myocardial infarction, stroke), major and minor bleeding, and death.

ELIGIBILITY:
Inclusion Criteria:

* with osteoarthritis
* scheduled for elective primary unilateral THR or TKR
* provided informed consent
* can read, write and speak English

Exclusion Criteria:

* history of arterial or venous thromboembolic disease (myocardial infarction, symptomatic ischemic heart disease, atrial fibrillation, cerebrovascular accident, deep-vein thrombosis, pulmonary embolus, or thrombogenic cardiac valvular disease or rhythm disease)
* pre-operative Hg of <120 g/L
* Known allergy to Tranexamic Acid
* Coagulation disorder
* Acquired disturbances of color vision
* Hepatic insufficiency, any history of liver disease
* Renal insufficiency (on dialysis)
* Preoperative prophylactic use of antiplatelet or anticoagulant therapy such as Clopidogrel, Warfarin, dabigatran or Rivaroxaban. This does not include low dose Aspirin (81mg)
* Patients with a history of subarachnoid hemorrhage [20]
* Simultaneous bilateral THA or TKA
* Any contra-indication for spinal anesthesia
* Allergy to Celecoxib, which will be the only nonsteroidal anti-inflammatory drugs (NSAID) used in the multi-modal analgesia regime.
* Retinal vein or retinal artery occlusion
* Female on oral contraceptive pills and/or premenopausal
* Concurrently taking hydrochlorothiazide, desmopressin, sulbactam-ampicillin, carbazochrome, ranitidine and/or nitroglycerin for the duration of the surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in hemoglobin during hospital stay | routinely measured post-op day 1 and 3

SECONDARY OUTCOMES:
Serum Troponin | Every 6 hours for 24 hours post-op
D-dimer | Post-op day 1 and 2

OTHER OUTCOMES:
Post-operative blood transfusion | During the first 7 days
  documentation of blood transfusion post-operative
Major or minor bleeding events | within 90 days of surgery
Self-reported visual disturbances | within 90 days of surgery
Self-reported symptomatic DVT | within 90 days of surgery
Self-reported PE | within 90 days of surgery
Self-reported stroke | within 90 days of surgery
Death | within 90 days of surgery
Intra-operative fluid balance | during surgery
  documentation of the volume of saline fluid via intravenous given to patients
Bleeding sources other than the knee or hip (eg: GI bleed) | within 90 days of surgery
post-operative fluid balance | within 3- 5 days of surgery
  documentation of the volume of saline fluid via intravenous given to patients

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Turgeon, MD, Principal Investigator — Concordia Joint Replacement Group
Locations (1):
- Concordia Hospital, Winnipeg, Manitoba, Canada